CLINICAL TRIAL: NCT04403854
Title: The ME-SH (Myalgic Encephalomyelitis in Stockholm-Harvard) Study: Structural Problems in Brainstem and Cervical Spine Cord in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome(ME/CFS) - a Case-control Study
Brief Title: Structural Problems in Brainstem and Cervical Spine Cord in ME/CFS
Status: Not yet recruiting | Type: Observational
Sponsor: Bragee Clinics (Other)
Responsible Party: Sponsor
Other Study IDs: BRAGEE MEPRO
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ME/CFS patients: Patients diagnosed according to Canada Criteria 2003
  Interventions: Diagnostic Test: MRI; Procedure: Spinal Tap
- Healthy Controls: Age and sex matched healthy controls
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — If possible with spectroscopy
  Other Names: Cervical MRI, Brain MRI
Procedure: Spinal Tap — together with CSF pressure estimate
  Other Names: CFS sampling
  Groups: ME/CFS patients

SUMMARY:
A case control study on patients with ME/CFS and healthy controls on prevalence of cervical obstructions, Cerebro spinal fluid (CSF) pressure and laboratory findings.

DETAILED DESCRIPTION:
50 patients and 50 healthy controls will undergo clinical exams and blood test of inflammatory and other findings as well as magnetic resonance imaging (MRI) with spectroscopy. The patients will undergo csf -sampling and measurements of CSF pressure.

ELIGIBILITY:
Inclusion Criteria:

Diagnose Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) according to Canada Consensus Criteria from 2003

Exclusion Criteria:

Bleeding abnormality Contraindication to Magnetic Resonance Imaging MRI Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnoses with ME/CFS and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalance of cervical obstructions | Two days
  MRI findings
Prevalence of Intracranial Hypertension | Two days
  CSF measurements

CONTACTS AND LOCATIONS:
Overall Officials: Björn Bragee, MD, Study Chair — Medect Clinical Trials

IPD SHARING:
Plan to Share IPD: Yes
Will be shared to other researchers with ethical approvement
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completed study or published results and 3 years thereafter
Access Criteria: Researchers with that have ethical approvement.
URL: http://www.bragee.se/research